CLINICAL TRIAL: NCT06717737
Title: Impact of Team-Based Training on Compliance and Physical Fitness in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shen Xin (Other)
Responsible Party: Sponsor-Investigator, Shen Xin, doctor, Hunan Normal University
Organization: Hunan Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20241225
Record Dates: First submitted 2024-10-29; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Physical Fitness Deficits in Firefighters; Exercise Adherence Challenges; Injury Risk Associated with Firefighting Tasks
Keywords: Team-Based Training; Firefighters; Physical Fitness; Exercise Adherence; Health Outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Team-Based Training Intervention for Firefighter Fitness and Adherence (Experimental): This arm involves a six-month team-based training intervention designed to improve firefighters' physical fitness and exercise adherence. The program includes aerobic, resistance, and functional exercises tailored to the demands of firefighting tasks. Sessions are conducted in small groups to foster teamwork and peer support, with participants receiving real-time feedback and guidance from certified professionals. The aim is to enhance cardiovascular fitness, strength, endurance, and overall health behaviors, while reducing injury risks. Participants track their progress using the Gymsmart (Pro X) app to monitor activity levels and adjust intensity for optimal results.
  Interventions: Behavioral: Intervention group：Conducted a 6-month team training intervention
- Control group (Experimental): The control group maintained their old habits
  Interventions: Behavioral: Control group： Maintaining old exercise habits

INTERVENTIONS:
Behavioral: Control group： Maintaining old exercise habits — The control group will maintain their original daily habits without any intervention behaviors for them
  Arms: Control group
Behavioral: Intervention group：Conducted a 6-month team training intervention — Spanning six months, the program incorporated aerobic training, resistance training, and functional exercises essential for rescue operations. Each training session was led by certified professionals who emphasized adherence to safety protocols and provided real-time feedback.
  Central to the training process was the significance of teamwork and mutual support, with sessions conducted in small groups focused on shared objectives. This framework fostered a collaborative environment that promoted peer support and motivated participants to actively engage in their fitness regimen. The group setting enabled firefighters to encourage one another and share individual progress, thereby enhancing their sense of responsibility and belonging.
  Arms: Team-Based Training Intervention for Firefighter Fitness and Adherence

SUMMARY:
Research Objectives: This study aims to develop a team-based training model specifically tailored for firefighters, focusing on improving their cardiovascular fitness, physical attributes, and fostering sustainable health behaviors. The ultimate goal is to reduce the risk of injuries associated with the physically demanding tasks they perform during their duties.

Research Hypotheses:

Firefighters participating in the team-based training model will demonstrate significant improvements in key fitness parameters, such as cardiorespiratory fitness, muscular strength, endurance, and body composition compared to those engaged in traditional training.

The team-based approach will enhance adherence to physical training among firefighters, leading to more consistent participation and improved health outcomes.

This clinical study is a randomized controlled trial that involved 42 firefighters who were divided into two groups: one receiving a team-based training intervention for six months and the other continuing with conventional exercises. The team training incorporated aerobic, resistance, and functional exercises, emphasizing teamwork and peer support to motivate participants. Key fitness measures, including cardiorespiratory fitness, strength, endurance, flexibility, and body mass index (BMI), were assessed before and after the intervention.

The study hypothesized that the team-based training model would not only enhance fitness levels but also improve adherence to training routines among firefighters, ultimately contributing to better health and safety during their demanding work.

ELIGIBILITY:
Inclusion Criteria:

Firefighters aged 18 to 50 years. Currently active duty within the selected brigade. Capable of performing physically demanding tasks without medical restrictions. Written informed consent provided by participants.

Exclusion Criteria:

Firefighters with any cardiovascular, respiratory, or musculoskeletal conditions that could hinder participation or affect fitness outcomes.

Individuals recovering from recent injuries or surgeries. Firefighters enrolled in external training programs that may impact baseline health assessments.

Any participant who refuses to provide informed consent.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max) | Baseline, 3 months, and 6 months following the intervention.
  This primary outcome measure assesses changes in cardiorespiratory fitness among firefighters participating in the team-based training program. Fitness is evaluated using the Gerkin treadmill protocol, which estimates maximal oxygen consumption (VO2max).
Body composition | Baseline, 3 months, and 6 months following the intervention.
  measured using the Inbody770 bioelectrical impedance analyzer, with BMI calculated as weight (kg) divided by height squared (m²);
Muscular strength | Baseline, 3 months, and 6 months following the intervention.
  Grip strength is assessed using a hand dynamometer, with the maximum value recorded from three attempts for each hand.
Muscular endurance | Baseline, 3 months, and 6 months following the intervention.
  Muscular endurance is evaluated through maximum push-ups and sit-ups performed within standardized time limits (2 minutes for push-ups and 3 minutes for sit-ups).
Flexibility | Baseline, 3 months, and 6 months following the intervention.
  Flexibility is assessed using a modified sit-and-reach test, measuring the distance reached beyond the toes while seated.
Exercise adherence | Baseline, 3 months, and 6 months following the intervention.
  Adherence is assessed by tracking the completion of daily training sessions, defined as performing more than 50% of the prescribed exercises and sets.

CONTACTS AND LOCATIONS:
Locations (1):
- Changsha Fire Brigade, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol